CLINICAL TRIAL: NCT00131768
Title: A Study of the Safety and Efficacy of Synvisc in Patients With Symptomatic Ankle Osteoarthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Medical Monitor, Genzyme Corporation
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYNV-003-02
Record Dates: First submitted 2005-08-17; First posted 2005-08-19 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Osteoarthritis
Keywords: osteoarthritis of the ankle; musculoskeletal
MeSH Terms: conditions — Osteoarthritis

INTERVENTIONS:
Device: Synvisc (hylan G-F 20)

SUMMARY:
This clinical study is to evaluate the safety and efficacy of Synvisc in patients with symptomatic ankle osteoarthritis (OA). Patients will be given Synvisc, with the possible administration of a second injection where insufficient symptomatic pain relief was experienced during the initial 3 months follow up period.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic OA pain of ankle (talo-crural)

Exclusion Criteria:

* Patients with current or prior conditions or treatments that would impede measurements of efficacy or safety

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-11; Study Completion 2006-02

PRIMARY OUTCOMES:
Pain relief

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (5):
- Germany (2):
  - Sportmedizinisches Institut Frankfurt am Main e.V. Orthopadie, Frankfurt
  - Johanna Etienne Krankenhaus, Neuss
- Italy (2):
  - Instituti Ortopedici Rizzoli, Bologna
  - Ospedale Santa Chiara, Clinica Ortopedica, Universita di Pisa, Pisa
- Academisch Medisch Centrum, Amsterdam, Netherlands